CLINICAL TRIAL: NCT01453387
Title: A Phase I Dose-Escalation First-In-Human Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Oral MEK Inhibitor MSC2015103B Administered With Two Different Treatment Schedules in Subjects With Advanced Solid Tumors
Brief Title: MSC2015103B in Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to an administrative reason
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200064-001
Record Dates: First submitted 2011-09-09; First posted 2011-10-17 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Advanced Solid Tumor
Keywords: MEK inhibitor; Solid Tumor; Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 - MSC2015103B (Schedule 1) (Experimental)
  Interventions: Drug: MSC2015103B
- Part 1 - MSC2015103B (Schedule 2) (Experimental)
  Interventions: Drug: MSC2015103B

INTERVENTIONS:
Drug: MSC2015103B — Schedule 1: MSC2015103B will be administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle until MTD establishment. Starting dose will be 150 microgram (mcg), which will be escalated to 200 mcg, 300 mcg, 450 mcg, 650 mcg, 1000 mcg and 1500 mcg subsequently.
  Arms: Part 1 - MSC2015103B (Schedule 1)
Drug: MSC2015103B — Schedule 2: MSC2015103B will be administered orally thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle until MTD was established. Starting dose will be 150 mcg, and will be escalated to 200 mcg subsequently.
  Arms: Part 1 - MSC2015103B (Schedule 2)

SUMMARY:
The main purpose of this study is to test the experimental drug, MSC2015103B at different dose levels and on different treatment schedules, to see whether it is safe and can be tolerated when given to subjects once a day one day per week over a 21-day period or once a day three times per week over a 21-day period. The investigators would also like to find out how MSC2015103B is broken down by the body.

Additional purposes of the trial are to assess side effects of MSC2015103B and to find out whether MSC2015103B has anti-cancer effects. In addition, the investigators would like to explore pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed solid tumor preferably, but not exclusively, including pancreatic, thyroid, colorectal, non-small cell lung, endometrial, renal, breast, ovarian carcinoma, or melanoma which is locally advanced or metastatic, and either refractory after standard therapy for the disease or for which no effective standard therapy is available
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of less than or equal to (<=) 1
* Has read and understands the informed consent form and is willing and able to give informed consent. Fully understands requirements of and willing to comply with all trial visits and assessments
* Evidence of measurable disease at trial entry as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.0.
* Willing to provide archival tissue samples for molecular analysis

Other inclusion criteria as defined in protocol.

Exclusion Criteria

* Bone marrow impairment as evidenced by hemoglobin less than (<) 9.0 gram per deciliter (g/dL), neutrophil count < 1.5 x 10^9 per liter (/L), and/or platelets <100 x 10^9/L per liter (/L)
* Renal impairment as evidenced by serum creatinine greater than (>) 1.5 x upper limit of normal (ULN) and/or calculated creatinine clearance < 50 milliliter per minute (mL/min) (Cockcroft-Gault formula)
* Liver function and liver cell integrity abnormality as defined by total bilirubin > 1.5 x ULN, or aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 2.5 x ULN, for subjects with liver involvement AST/ALT > 5 x ULN. Subjects with albumin < 2.5 g/dL are also excluded
* History of central nervous system (CNS) metastases.
* History of difficulty of swallowing, malabsorption, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the tested product.
* Chronic diarrhea that is >= Grade 2 in severity
* Clinically significant cardiac conduction abnormalities
* A left ventricular ejection fraction of < 45%
* A history of stroke or myocardial infarction within the past year
* A history of uveitis and scleritis
* Retinal pathology beyond normal age-related processes
* Evidence of a retinal vein occlusion on fluorescein angiogram or a history of retinal vein occlusion
* Subjects are also excluded if their ophthalmologist finds that their optic disc is at risk for a central retinal vein occlusion
* History of glaucoma
* Subjects requiring daily and/or chronic systemic steroids
* Pregnant or nursing females Other exclusion criteria as defined in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono, a division of Merck KGaA, Darmstadt, Germany
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): 09 September 2011/18 April 2013. Study completion date: 15 July 2013, Clinical data cut-off date: 15 July 2013; Subjects were randomized at 3 centers in United States.
Pre-assignment Details: Enrolled: 28 subjects were screened for eligibility and all were randomized in to the trial.
Groups:
- Part 1 - MSC2015103B (Schedule 1): MSC2015103B was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle until maximum tolerated dose (MTD) was established. Starting dose was 150 microgram (mcg), which was escalated to 200 mcg, 300 mcg, 450 mcg, 650 mcg, 1000 mcg and 1500 mcg subsequently.
- Part 1 - MSC2015103B (Schedule 2): MSC2015103B was administered orally thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle until MTD was established. Starting dose was 150 mcg, and was escalated to 200 mcg subsequently.
Period: Overall Study
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Started | 21 | 7
Completed | 21 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least one administration of the trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2) | Total
Number analyzed (Participants) | 21 | 7 | 28
Age, Customized [Number; unit: Subjects]
  18 to less than (<) 45 years | 2 | 0 | 2
  Greater than equal to (>=) 45 to <65 years | 10 | 5 | 15
  >=65 years | 9 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 17 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Dose-limiting Toxicities (DLT)
Description: DLT was evaluated using the National cancer institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. DLT was defined as any of the following AEs occurring during Cycle 1 that are not related to progressive disease (PD) at any dose level: Any Grade 3 or more non-hematological toxicity excluding: Grade 3 diarrhea or associated electrolyte abnormalities that were controlled with adequate and optimal therapies, Grade 3 liver function abnormalities which resolved within 7 days, vomiting. Grade 4 neutropenia of greater than (>) 5 days duration or Grade 3 febrile neutropenia, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding, any severe or life threatening AE or any AE or abnormality which impairs daily normal physiological functions, any treatment delay for 2 weeks or more due to adverse effects not related to PD. All events judged to be related by the Investigator to PD were excluded from the DLT definition.
Time Frame: Up to Day 21 of Cycle 1
Population: Safety analysis set included all the subjects who received at least one administration of the trial medication.
Measure: Number; unit: Subjects
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
Subjects | 0 | 0

2. Primary Outcome: Percentage of Subjects Who Experienced DLT
Description: DLT was evaluated using the National cancer institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. DLT was defined as any of the following AEs occurring during Cycle 1 that are not related to PD at any dose level: Any Grade 3 or more non-hematological toxicity excluding: Grade 3 diarrhea or associated electrolyte abnormalities that were controlled with adequate and optimal therapies, Grade 3 liver function abnormalities which resolved within 7 days, vomiting. Grade 4 neutropenia of greater than (>) 5 days duration or Grade 3 febrile neutropenia, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding, any severe or life threatening AE or any AE or abnormality which impairs daily normal physiological functions, any treatment delay for 2 weeks or more due to adverse effects not related to PD. All events judged to be related by the Investigator to PD were excluded from the DLT definition.
Time Frame: Up to Day 21 of Cycle 1
Population: Safety analysis set included all subjects who received at least one administration of the trial medication.
Measure: Number; unit: Percentage of subjects
Groups:
- Part 1 - MSC2015103B (Schedule 1): MSC2015103B was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle until MTD was established. Starting dose was 150 microgram (mcg), which was escalated to 200 mcg, 300 mcg, 450 mcg, 650 mcg, 1000 mcg and 1500 mcg subsequently.
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
Percentage of subjects | 0 | 0

3. Secondary Outcome: Percentage of Subjects Who Experienced Any Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death and TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. SAE (Serious adverse event) is defined as any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition.. TEAEs are events between first dose of study drug up to the cut-off date (15 July 2013) and were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the initiation of the trial till the data cut-off date 15 July 2013
Population: The safety analysis set included all the subjects who received at least one administration of the trial medication.
Measure: Number; unit: Percentage of subjects
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
Percentage of subjects
  TEAEs | 100.0 | 100.0
  Serious TEAEs | 19.0 | 42.9
  TEAEs leading to death | 0.0 | 0.0
  TEAEs leading to discontinuation | 0.0 | 14.3

4. Secondary Outcome: Percentage of Subjects Who Experienced Clinically Significant Lab Abnormality Judged to be Related to the Trial Medication
Description: Abnormal laboratory findings and other abnormal investigational findings which were associated with clinical signs and symptoms, lead to treatment discontinuation, or considered medically important by the investigator were reported as AEs.
Time Frame: From the initiation of the trial till the data cut-off date 15 July 2013
Population: The safety analysis set included all the subjects who received at least one administration of the trial medication.
Measure: Number; unit: Percentage of subjects
Groups:
- Part 1 - MSC2015103B 200 mcg (Schedule 1): The planned dose of MSC2015103B (150 mcg, 200 mcg, 300 mcg, 450 mcg, 650 mcg, 1000 mcg and 1500 mcg) was orally administered once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B (Schedule 2): The planned dose of MSC2015103B (150 mcg and 200 mcg) was orally administered thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle.
Arm/Group | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
Percentage of subjects
  Aspartate aminotransferase increased | 14.3 | 0.0
  Decreased appetite | 14.3 | 14.3
  Gamma-glutamyl transferase increased | 0.0 | 14.3
  Blood alkaline phosphatase increased | 0.0 | 14.3
  Ejection fraction decreased | 0.0 | 14.3
  Blood glucose increased | 0.0 | 14.3
  Hypokalemia | 0.0 | 28.6
  Hyponatraemia | 0.0 | 28.6
  Hypoalbuminaemia | 0.0 | 14.3
  Hypophosphatemia | 0.0 | 14.3

5. Secondary Outcome: Number of Subjects Who Experienced Clinically Significant Lab Abnormality Judged to be Related to the Trial Medication
Description: as for outcome 4
Time Frame: From the initiation of the trial till the data cut-off date 15 July 2013
Population: The safety analysis set included all the subjects who received at least one administration of the trial medication.
Measure: Number; unit: Subjects
Groups:
- Part 1 - MSC2015103B (Schedule 1): The planned dose of MSC2015103B (150 mcg, 200 mcg, 300 mcg, 450 mcg, 650 mcg, 1000 mcg and 1500 mcg) was orally administered once weekly on Days 1, 8, and 15 of a 21-day cycle.
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
Subjects
  Aspartate aminotransferase increased | 3 | 0
  Decreased appetite | 3 | 1
  Gamma-glutamyl transferase increased | 0 | 1
  Blood alkaline phosphatase increased | 0 | 1
  Ejection fraction decreased | 0 | 1
  Blood glucose increased | 0 | 1
  Hypokalemia | 0 | 2
  Hyponatraemia | 0 | 2
  Hypoalbuminaemia | 0 | 1
  Hypophosphatemia | 0 | 1

6. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: Schedule 1 : 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, 24.0, 48 or 72, 72 or 96 and 168 hours post-dose during Week 1 and Week 3; Schedule 2: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, and 24.0 hours post-dose on Days 1 and 17.
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of MSC2015103B and provided sufficient plasma concentrations of MSC2015103B measurement after the first dose. "n" signifies the number of subjects evaluable for the particular timepoint.
Measure: Geometric Mean (Full Range); unit: Picogram per milliliter
Groups:
- Part 1 - MSC2015103B 150 mcg (Schedule 1): MSC2015103B 150 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 200 mcg (Schedule 1): MSC2015103B 200 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 300 mcg (Schedule 1): MSC2015103B 300 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 450 mcg (Schedule 1): MSC2015103B 450 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 650 mcg (Schedule 1): MSC2015103B 650 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 1000 mcg (Schedule 1): MSC2015103B 1000 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 1500 mcg (Schedule 1): MSC2015103B 1500 mcg was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle.
- Part 1 - MSC2015103B 150 mcg (Schedule 2): MSC2015103B 150 mcg was administered orally thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle.
- Part 1 - MSC2015103B 200 mcg (Schedule 2): MSC2015103B 200 mcg was administered orally thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle.
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
Picogram per milliliter
  Week 1 (n=3, 4, 3, 3, 3, 3, 2, 3, 4) | 38.750 [25.20 to 58.90] | 38.110 [25.40 to 56.70] | 97.293 [34.40 to 179.2] | 290.98 [199.1 to 441.0] | 396.45 [193.7 to 657.2] | 888.15 [295.0 to 3010] | 2215.9 [1760 to 2790] | 75.313 [55.60 to 98.50] | 52.331 [33.4 to 72.7]
  Week 2 (n= 3,3,3,3,1,3,2,2,3) | 48.952 [29.70 to 82.80] | 63.732 [54.50 to 74.80] | 219.71 [108.1 to 336.1] | 329.62 [257.3 to 439.5] | 2471.0 [2471 to 2471] | 1728.1 [835.0 to 2630] | 5636.8 [5340 to 5950] | 190.59 [141.4 to 256.9] | 157.62 [80.10 to 404.0]

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: Schedule 1: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, 24.0, 48 or 72, 72 or 96 and 168 hours post-dose during Week 1 and Week 3; Schedule 2: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, and 24.0 hours post-dose on Day 1 and 17.
Population: as for outcome 6
Measure: Geometric Mean (Full Range); unit: Hour
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
Hour
  Week 1 (n=3,4,3,3,3,3,2,3,4) | 2.4478 [1.833 to 4.000] | 5.2643 [4.000 to 8.000] | 1.4422 [1.000 to 2.000] | 1.4422 [1.000 to 2.000] | 1.5874 [1.000 to 4.0000] | 1.1447 [0.500 to 2.000] | 1.2450 [1.033 to 1.500] | 2.4248 [1.500 to 6.067] | 1.3161 [1.000 to 2.000]
  Week 3 (n=3,3,3,3,1,3,2,2,3) | 1.1573 [1.000 to 1.500] | 2.3833 [1.500 to 6.017] | 4.5789 [2.000 to 8.000] | 1.1635 [1.000 to 1.500] | 0.50000 [0.5000 to 0.5000] | 2.0110 [1.017 to 4.000] | 0.70711 [0.5000 to 1.000] | 2.8519 [2.033 to 4.000] | 1.6869 [1.500 to 2.133]

8. Secondary Outcome: Apparent Terminal Half Life (T1/2)
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50% in the final stage of its elimination.
Time Frame: as for outcome 7
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of MSC2015103B and provided sufficient plasma concentrations of MSC2015103B measurement after the first dose."n" signifies the number of subjects evaluable for the particular timepoint.
Measure: Geometric Mean (Full Range); unit: Hour
Groups:
- Part 1 - MSC2015103B 200 mcg (Schedule 2): MSC2015103B 200 mcg was orally administered thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle.
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
Hour
  Week 1 (n=3,4,3,3,3,3,2,3,4) | 134.88 [72.76 to 201.9] | 115.41 [73.51 to 280.2] | 55.023 [20.85 to 118.7] | 53.072 [51.51 to 55.10] | 115.34 [85.23 to 135.4] | 52.852 [49.40 to 58.26] | 81.124 [33.51 to 196.4] | 30.850 [23.55 to 40.09] | 33.007 [22.74 to 46.98]
  Week 3 (n=3,3,3,3,1,3,2,2,3) | 102.30 [41.27 to 251.3] | 102.53 [76.49 to 122.5] | 138.47 [115.5 to 191.1] | 55.43 [42.21 to 85.54] | 37.16 [37.16 to 37.16] | 103.77 [55.95 to 185.7] | 100.91 [91.41 to 111.4] | 121.58 [49.19 to 300.5] | 145.70 [56.03 to 643.5]

9. Secondary Outcome: Area Under the Plasma Concentration Curve From Time Zero to Infinity (AUC[0-inf])
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: as for outcome 7
Population: Pharmacokinetic analysis set included all the subjects who have received at least 1 dose of MSC2015103B and provided sufficient plasma concentrations of MSC2015103B measurement after the first dose. "n" signifies the number of subjects evaluable for the particular timepoint.
Measure: Geometric Mean (Full Range); unit: Hour*picogram/milliliter
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
Hour*picogram/milliliter
  Week 1 (n=3,4,3,3,3,3,2,3,4) | 3644.7 [1997 to 6477] | 3927.4 [2513 to 5479] | 2249.9 [829.0 to 4037] | 7890.1 [6454 to 10920] | 12454 [8921 to 23730] | 13164 [6049 to 19880] | 23558 [18580 to 29870] | 2032.2 [1408 to 3234] | 1375.2 [948.0 to 2377]
  Week 3 (n=,3,3,3,3,1,3,2,2,3) | 4715.2 [1710 to 17490] | 4377.2 [3552 to 6006] | 16465 [7797 to 38300] | 12397 [7532 to 16750] | 24580 [24580 to 24580] | 35423 [14410 to 68400] | 66081 [61480 to 71020] | 21735 [6093 to 77530] | 14870 [7409 to 27350]

10. Secondary Outcome: AUC Versus Time Curve Within One Dosing Interval (AUC0-tau)
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Full Range); unit: hours*picogram/milliliter
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
hours*picogram/milliliter
  Week 1 (n=3,4,3,3,3,3,2,3,4) | 2072.8 [1549 to 2789] | 2381.6 [1947 to 3892] | 1752.7 [725.1 to 3202] | 6824.4 [5577 to 9363] | 8434.6 [6120 to 13990] | 11533 [5498 to 17850] | 17698 [16630 to 18830] | 1345.3 [1073 to 1809] | 865.76 [738.5 to 1231]
  Week 3 (n=3,3,3,3,1,3,2,2,3) | 2946.9 [1645 to 6147] | 3002.0 [2525 to 3810] | 8865.3 [4920 to 16490] | 10696 [7208 to 15580] | 23670 [23670 to 23670] | 25150 [12190 to 40520] | 47114 [44670 to 49690] | 4993.3 [2984 to 8356] | 3070.5 [1661 to 7338]

11. Secondary Outcome: Apparent Oral Clearance of the Drug From Plasma (CL/f)
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/f was influenced by the fraction absorbed.
Time Frame: Schedule 1: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, 24.0, 48 or 72, 72 or 96 and 168 hours post-dose during Week 1; Schedule 2: 0, 0.5, 1.0, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, and 24.0 hours post-dose on Day 1.
Population: Pharmacokinetic analysis set included all the subjects who have received at least one dose of MSC2015103B and who have provided sufficient plasma concentrations of MSC2015103B measurement after the first dose. "N" signifies the total number of subjects evaluable for this outcome measure.
Measure: Geometric Mean (Full Range); unit: Liter/hour
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
Liter/hour | 41.156 [23.16 to 75.11] | 50.924 [36.51 to 79.57] | 133.34 [74.30 to 361.9] | 57.033 [41.19 to 69.73] | 52.192 [27.39 to 72.86] | 75.968 [50.29 to 165.3] | 63.673 [50.22 to 80.73] | 73.813 [46.38 to 106.6] | 145.44 [84.15 to 211.0]

12. Secondary Outcome: Apparent Volume of Distribution Associated to the Terminal Phase (Vz/f)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed.
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of MSC2015103B and who provided sufficient plasma concentrations of MSC2015103B measurement after the first dose. "n" signifies the number of subjects evaluable for the particular timepoint.
Measure: Geometric Mean (Full Range); unit: Liter
Groups:
- Part 1 - MSC2015103B 150 mcg (Schedule 2): MSC2015103B 150 mcg was orally administered thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle.
Arm/Group | Part 1 - MSC2015103B 150 mcg (Schedule 1) | Part 1 - MSC2015103B 200 mcg (Schedule 1) | Part 1 - MSC2015103B 300 mcg (Schedule 1) | Part 1 - MSC2015103B 450 mcg (Schedule 1) | Part 1 - MSC2015103B 650 mcg (Schedule 1) | Part 1 - MSC2015103B 1000 mcg (Schedule 1) | Part 1 - MSC2015103B 1500 mcg (Schedule 1) | Part 1 - MSC2015103B 150 mcg (Schedule 2) | Part 1 - MSC2015103B 200 mcg (Schedule 2)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 2 | 3 | 4
Liter | 8008.6 [6746 to 9658] | 8478.7 [4275 to 14760] | 10584 [7219 to 15090] | 4366.9 [3275 to 5298] | 8684.7 [5349 to 13670] | 5792.4 [3722 to 11780] | 7452.2 [3903 to 14230] | 3285.2 [2682 to 3651] | 6925.6 [5704 to 8253]

13. Secondary Outcome: Extracellular Signal-regulated Kinase (ERK) Phosphorylation Levels
Description: ERK phosphorylation levels were to be assessed in peripheral blood mononuclear cells (PBMC) during the dose escalation
Time Frame: Schedule 1: Day 1: Pre-dose; Post-dose: 2, 4, 8, 24 hour; 48 or 72 hour; 48 or 96 hour, 168 hour; Day 15: Pre-dose; Schedule 2: Day 1: Pre-dose; Post-dose: 2, 8, 24, 48, 96 hour; Day 15: Pre-dose; Day 17: Pre-dose; Post-dose: 2, 8, and 24 hour
Population: As the trial was terminated early due to administrative reason, it was decided as per Statistical Analysis Plan not to evaluate the biomarker data for this study.
Groups:
- Part 1 - MSC2015103B (Schedule 1): MSC2015103B was administered orally once weekly on Days 1, 8, and 15 of a 21-day cycle until MTD was established. Starting dose was 150 mcg, which was escalated to 200 mcg, 300 mcg, 450 mcg, 650 mcg, 1000 mcg and 1500 mcg.
- Part 1 - MSC2015103B (Schedule 2): MSC2015103B was administered orally thrice weekly on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19 of a 21-day cycle until MTD was established. Starting dose was 150 mcg, which was escalated to 200 mcg.
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Subjects With Overall Response
Description: Overall response was to be confirmed by complete response (CR) or partial response (PR) using response evaluation criteria in solid tumours Version 1.0 (RECIST) during treatment. CR: The disappearance of all target and non-target lesions and normalization of tumor marker level; PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the sum of the longest diameter at baseline.
Time Frame: Every 6 Weeks until complete response or till data cut-off date 15 July 2013
Population: The efficacy analysis set included all subjects who received at least 1(non-zero) dose of MSC2015103B and had a baseline tumor assessment.
Measure: Number; unit: percentage of subjects
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
percentage of subjects
  CR | 0 | 0
  PR | 0 | 0

15. Secondary Outcome: Percentage of Subjects With Clinical Benefit
Description: Clinical benefit was to be confirmed by CR, PR or stable disease (SD) lasting at least 6 weeks (using RECIST v1.0) during treatment. CR: The disappearance of all target and non-target lesions and normalization of tumor marker level; PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the sum of the longest diameter at baseline; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since treatment started.
Time Frame: Every 6 Weeks until complete response or till data cut-off date 15 July 2013
Population: as for outcome 14
Measure: Number; unit: percentage of subjects
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Number analyzed (Participants) | 21 | 7
percentage of subjects | 33.3 | 28.6

ADVERSE EVENTS:
Time Frame: From the initiation of the trial till data cut-off date (15 July 2013)
Arm/Group | Part 1 - MSC2015103B (Schedule 1) | Part 1 - MSC2015103B (Schedule 2)
Serious Adverse Events (participants affected / at risk) | 4/21 | 3/7
Other Adverse Events (participants affected / at risk) | 21/21 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - MSC2015103B (Schedule 1) (N=21) | Part 1 - MSC2015103B (Schedule 2) (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - MSC2015103B (Schedule 1) (N=21) | Part 1 - MSC2015103B (Schedule 2) (N=7)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve sclerosis (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Retching (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Axillary pain (General disorders) | 1 | 0
Breakthrough pain (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Early satiety (General disorders) | 1 | 1
Fatigue (General disorders) | 9 | 2
Influenza like illness (General disorders) | 1 | 1
oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 1 | 2
Device occlusion (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0
Breathe sounds abnormal (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 1
Gamma-glutamyl transferase increased (Investigations) | 4 | 1
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Protein total increased (Investigations) | 1 | 0
Weight increased (Investigations) | 4 | 0
Blood glucose increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Backpain (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hydroureter (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Biliary drainage (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early during Part 1 of the trial due to administrative reason. Pharmacodynamics evaluations were not performed due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study as a whole will be published prior to any individual investigator publications. It is required that copies of all papers, abstracts, articles, etc. that contain study data are to be forward to the Sponsor for review 30 days prior to submission for publication.